CLINICAL TRIAL: NCT04442152
Title: Phone Survey for Understanding the Impact of COVID-19 on Caregiving and Family Dynamics on Bandebereho Study Participants
Brief Title: Impact of COVID-19 on Family Dynamics on Bandebereho Study Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Promundo, United States (Other)
Collaborators: Rwanda Men's Resource Center (Rwamrec) (Unknown); Ministry of Health/Rwanda Biomedical Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 265A
Record Dates: First submitted 2020-06-19; First posted 2020-06-22 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Gender Relations; Partner Communication; Division of Carework; Couple Conflict; Stress
Keywords: gender, caregiving, Covid-19, couple relations
MeSH Terms: conditions — Coitus; COVID-19

STUDY DESIGN:
Intervention Model Description: Note that we are collecting new data from participants previously randomly assigned to intervention and control arms.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): See intervention description
  Interventions: Behavioral: MenCare+/Bandebereho fathers'/couples' group education
- Control (No Intervention): Participants who were randomized into the control arm were and will be surveyed at the same time point as intervention participants, but did not receive any intervention.

INTERVENTIONS:
Behavioral: MenCare+/Bandebereho fathers'/couples' group education — MenCare+/Bandebereho is a 3 year project to engage men in maternal, newborn and child health (MNCH) and in sexual and reproductive health in Rwanda. A core component of the project is fathers'/couples' group education. The target participants were first-time parents or parents of young children living in 16 rural and semi-urban sectors selected by the implementing partner in collaboration with local authorities. The MenCare+/Bandebereho fathers'/couples' group education engages men in 15 weekly sessions of group discussion, critical reflection and interactive activities led by a trained facilitator using a curriculum developed by RWAMREC and Promundo and approved by the Rwandan Ministry of Health, adapted from the Program P Manual. Men's partners participate in 6-8 sessions. The sessions focus on men's role in MNCH, family planning, sharing household responsibilities, intimate partner violence, conflict resolution, family budgeting, and gender equality.
  Other Names: Program P
  Arms: Intervention

SUMMARY:
This proposed study will assess how COVID-19 and the associated 'stay at home' orders are affecting low-income Rwandan couples' relationships and family dynamics. The study builds on an existing randomized controlled trial of the Bandebereho fathers/couples intervention (NCT02694627), which will allow us to assess not only the current conditions in households, but also whether or how the significant impacts of the intervention are sustained under extreme stress.

DETAILED DESCRIPTION:
This proposed study will assess how COVID-19 and the associated 'stay at home' orders are affecting low-income Rwandan couples' relationships and family dynamics. It will contribute to documenting whether and how this disruptive moment might be changing or influencing relationship dynamics, conflict, and the distribution of care-work. We will build on an existing randomized controlled trial of the Bandebereho fathers/couples intervention, which will allow us to assess not only the current conditions in households, but also whether or how the significant impacts of the intervention are sustained under extreme stress. The Bandebereho fathers/couples intervention was implemented by the Rwanda Men's Resource Center (RWAMREC) and Promundo-US, in collaboration with the Rwanda Ministry of Health and local authorities in Karongi, Musanze, Nyaruguru and Rwamagana districts from 2013-2015. Results from a randomized controlled study of Bandebereho, a gender transformative intervention for expectant couples originally implemented in 4 districts in 2015, showed positive results across multiple outcomes after 21 months.

ELIGIBILITY:
Original inclusion criteria in the original RCT study included, for men: being between the ages of 21-35, expecting a child or having one or more children under the age of five, living in a stable partnership, and residing in the study site. For women, the criteria were simply being the partner of one of the men selected for the study.

Inclusion criteria for this study include previous participation in the RCT, and that the respondent indicated they or their partner owned a telephone/phone in the 21-month follow up that was conducted in November/December 2016. Based on data from the 21-month followup, approximately 80% of respondents reported a cell phone owned by them or their partner.

Ages: 26 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 998 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-09-04 (Actual)

PRIMARY OUTCOMES:
Gender division of caregiving/domestic tasks | ~5 years post intervention
  Question about how caregiving is distributed in the wake of Covid-19
Couple communication | ~5 years post intervention
  Frequency of couple communication in the wake of Covid-19
Couple conflict | ~5 years post intervention
  Frequency of couple quarreling in the wake of Covid-19
Men's alcohol use | ~5 years post intervention
  Frequency of men's alcohol use in the wake of Covid-19
Household economic situation | ~5 years post intervention
  Changes in household economic situation in the wake of Covid-19
Stress and frustration | ~5 years post intervention
  Feelings of stress and frustration in the wake of Covid-19

CONTACTS AND LOCATIONS:
Overall Officials: Kate E Doyle, MA, Principal Investigator — Promundo-US; Ruti G Levtov, PhD, Principal Investigator — Promundo-US; Felix Sayingoza, MD, MSc, Principal Investigator — Ministry of Health/Rwanda Biomedical Center; Fidele Rutayisire, MA, Principal Investigator — Rwanda Men's Resource Center; Shamsi Kazimbaya, MA, Principal Investigator — Promundo-US
Locations (1):
- Rwanda Men's Resource Centre (Rwamrec), Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doyle K, Levtov RG, Barker G, Bastian GG, Bingenheimer JB, Kazimbaya S, Nzabonimpa A, Pulerwitz J, Sayinzoga F, Sharma V, Shattuck D. Gender-transformative Bandebereho couples' intervention to promote male engagement in reproductive and maternal health and violence prevention in Rwanda: Findings from a randomized controlled trial. PLoS One. 2018 Apr 4;13(4):e0192756. doi: 10.1371/journal.pone.0192756. eCollection 2018. PMID 29617375